CLINICAL TRIAL: NCT05071664
Title: A Phase 2a, Multicenter, Randomized, Double-blind Study Evaluating the Efficacy and Safety of Subcutaneously Administered Guselkumab and Golimumab Combination Therapy in Participants With Active Psoriatic Arthritis
Brief Title: A Study of Guselkumab and Golimumab Combination Therapy in Participants With Active Psoriatic Arthritis
Acronym: AFFINITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109054; CNTO1959PSA2003 (Other: Janssen Research & Development, LLC); 2021-002012-31 (EudraCT Number)
Record Dates: First submitted 2021-09-06; First posted 2021-10-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab; golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Guselkumab and Golimumab (Experimental): Participants will receive subcutaneous (SC) guselkumab and golimumab.
  Interventions: Drug: Guselkumab; Drug: Golimumab
- Group 2: Guselkumab and Placebo (Active Comparator): Participants will receive SC guselkumab and placebo.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered as a SC injection.
  Other Names: TREMFYA; CNTO1959
Drug: Golimumab — Golimumab will be administered as a SC injection.
  Other Names: SIMPONI; CNTO148
  Arms: Group 1: Guselkumab and Golimumab
Drug: Placebo — Placebo will be administered as a SC injection.
  Arms: Group 2: Guselkumab and Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab plus golimumab combination treatment in participants with active psoriatic arthritis (PsA) and inadequate response (IR) to prior anti-tumor necrosis factor-alpha (anti-TNF-alpha) therapies by assessing clinical response compared with guselkumab monotherapy.

DETAILED DESCRIPTION:
PsA is a chronic inflammatory multi-faceted disease that impacts the peripheral and axial joints, soft tissues, and skin. Guselkumab is a fully human monoclonal antibody (mAb) directed against the p19 subunit of interleukin (IL)-23, blocks the binding of extracellular IL-23 to the cell surface IL-23 receptor, inhibiting IL-23 specific intracellular signaling, subsequent activation, and cytokine production. Golimumab is a fully human anti-TNF-alpha mAb that binds to TNF-alpha with high affinity, prevents binding to its receptors, thereby inhibiting the biological activity of TNF-alpha and resulting in limited production or activity of inflammatory cytokines, thereby providing therapeutic benefit in various chronic inflammatory disorders, including PsA. This study will consist of a Screening Phase (up to 6 weeks), Double-blind Phase from Weeks 0 to 24 which includes the active treatment phase and the primary efficacy visit (Week 24), and Safety Follow-up Phase from Week 24 to Week 36. Key safety assessments will include adverse events (AEs), clinical laboratory safety tests (hematology and chemistry), vital signs, monitoring for injection-site and hypersensitivity reactions, and early detection of active tuberculosis (TB). The total duration of the study is up to 42 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of psoriatic arthritis (PsA) for greater than or equal to (>=) 6 months prior to the first administration of study intervention and meet Classification criteria for PsA (CASPAR) criteria at screening
* Have active PsA as defined by having at least 3 swollen joints and at least 3 tender joints at screening and at baseline
* Have at least 1 of the following PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Have active plaque psoriasis, with at least one psoriatic plaque of >=2 centimeter (cm) diameter or nail changes consistent with psoriasis
* Have an inadequate response (IR) to anti-tumor necrosis factor-alpha (anti-TNF-alpha) therapy, defined as presence of active PsA despite treatment with either 1 or 2 prior anti-TNF-alpha agent(s) and the following: a. Lack of benefit to either 1 or 2 prior anti-TNF-alpha therapies, as documented in the participant history by the treating physician, after at least 12 weeks of etanercept, adalimumab, or certolizumab pegol therapy, or at least 14-weeks of infliximab, or any biosimilar of these 4 therapies. Documented lack of benefit may include inadequate improvement in joint counts, physical function, or disease activity; b. The last dose of anti-TNF-alpha therapy must have occurred greater than 5 half-lives of the drug prior to first study intervention administration (washout period)

Exclusion Criteria:

* Has other inflammatory diseases that might confound the evaluations of benefit of guselkumab and/or golimumab therapy, including but not limited to rheumatoid arthritis (RA), ankylosing spondylitis (AS), nonradiographic axial spondyloarthritis (nr AxSpA), systemic lupus erythematosus, or lyme disease
* Has known intolerance or hypersensitivity to any biologic medication, or known allergies or clinically significant reactions to murine, chimeric, or human proteins, monoclonal antibodies (mAb), or antibody fragments
* Has received prior treatment with golimumab or guselkumab or has documented intolerance to prior anti-TNF-alpha therapy in the participant history by the treating physician
* Has received more than 2 prior anti-TNF-alpha agents (or biosimilars)
* Positive human immunodeficiency virus (HIV) antibody test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Minimal Disease Activity (MDA) at Week 24 | Week 24
  MDA defines a satisfactory state of disease activity that includes the 5 domains of psoriatic arthritis (PsA; joint symptoms, skin psoriasis, participant's assessment of pain and disease activity, physical function, and enthesitis). Participants are classified as achieving MDA if they fulfilled 5 of 7 outcome measures: tender joint count less than or equal to (<=) 1; swollen joint count <=1; psoriasis area and severity index (PASI) <=1 or body surface area (BSA) <=3 percent (%); participant's pain visual analog scale (VAS) score of <=15; participant's global disease activity VAS (arthritis and psoriasis) score of <=20; disability index of the health assessment questionnaire (HAQ-DI) score <=0.5; and tender entheseal points <=1.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve American College of Rheumatology (ACR) 50 at Week 24 | Week 24
  ACR 50 response is defined as greater than or equal to (>=) 50% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints) and >=50% improvement from baseline in 3 of the following 5 assessments: participant's assessment of pain using VAS (0-100 millimeter [mm], 0 mm=no pain and 100 mm=worst possible pain), participant's global assessment of disease activity by using VAS (scale ranges from 0 mm to 100 mm, [0 mm= very well to 100 mm= very poor]), physician's global assessment of disease activity using VAS (scale ranges from 0 to 100, [0 = no arthritis to 100 = extremely active arthritis]), participant's assessment of physical function measured by HAQ-DI, defined as a 20-question instrument assessing 8 functional areas. The derived HAQ-DI ranges from 0 (indicating no difficulty), to 3 (indicating inability to perform a task in that area) and c-reactive protein (CRP).
Percentage of Participants who Achieve MDA at Week 16 | Week 16
  MDA defines a satisfactory state of disease activity that includes the 5 domains of PsA (joint symptoms, skin psoriasis, participant's assessment of pain and disease activity, physical function, and enthesitis). Participants are classified as achieving MDA if they fulfilled 5 of 7 outcome measures: tender joint count <=1; swollen joint count <=1; PASI <=1 or BSA <=3%; participant's pain VAS score of <=15; participant's global disease activity VAS (arthritis and psoriasis) score of <=20; HAQ-DI score <=0.5; and tender entheseal points <=1.
Percentage of Participants who Achieve PASI 90 at Week 24 Among the Participants with >=3% BSA Psoriatic involvement and an IGA Score of >=2 (Mild) at Baseline | Week 24
  The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. A PASI 90 response is defined as >=90% improvement in PASI score from baseline.
Percentage of Participants who Achieve PASI 100 at Week 24 Among the Participants with >=3% BSA Psoriatic involvement and an IGA Score of >=2 (Mild) at Baseline | Week 24
  The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. A PASI 100 response is defined as 100% improvement in PASI score from baseline.
Percentage of Participants with an IGA-psoriasis Response of IGA Psoriasis Score of 0 or 1 AND >=2 Grade Reduction From Baseline at Week 24 Among Participants with >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline | Week 24
  IGA psoriasis response is defined as an IGA psoriasis score of 0 (cleared) or 1 (minimal) and >=2 grade reduction from baseline. The IGA documents the investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling, each using a 5-point scale: using 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe) scale. The IGA score of psoriasis is based upon the average of induration, erythema, and scaling scores. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Change from Baseline in HAQ-DI at Week 24 | Baseline and Week 24
  HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3 where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning. Negative change from baseline indicates improvement of physical function.
Percentage of Participants With Resolution of Enthesitis at Week 24 Among the Participants With Enthesitis at Baseline | Week 24
  Enthesitis will be assessed using the Leeds Enthesitis Index (LEI), a tool developed to assess enthesitis in participants with PsA and evaluates the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The enthesitis index score is a total score of the 6 evaluated sites from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). A LEI score of 0 at a post baseline visit indicates resolution of enthesitis when baseline LEI >0.
Percentage of Participants with Resolution of Dactylitis at Week 24 Among the Participants with Dactylitis at Baseline | Week 24
  The presence and severity of dactylitis is assessed in both hands and feet using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. The results are summed to produce a final score ranging from 0 to 60. Higher score indicates more severe dactylitis. Resolution of dactylitis is defined as a dactylitis score of 0 with the baseline dactylitis score >0.
Change from Baseline in Short Form Health Survey (SF-36) Physical Component Score (PCS) at Week 24 | Baseline and Week 24
  SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a PCS with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The PCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Reasonably Related AEs | Up to 42 weeks
  Percentage of participants with AEs, SAEs, and reasonably related AEs will be assessed. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect, and suspects transmission of any infectious agent via a medicinal product. Reasonably related AEs are those AEs which are judged related to study treatment by the investigator.
Percentage of Participants With AEs Leading to Discontinuation of Study Intervention | Up to 42 weeks
  Percentage of participants with AEs leading to discontinuation of study intervention will be reported.
Percentage of Participants With Infections | Up to 42 weeks
  Percentage of participants with infections will be reported.
Percentage of Participants With Injection-site Reactions | Up to Week 20
  Percentage of participants with injection-site reactions will be reported. An injection-site reaction is any adverse reaction at a subcutaneous (SC) study intervention injection-site.
Serum Guselkumab and Golimumab Concentration | Up to Week 36
  Serum guselkumab and golimumab concentration will be measured.
Percentage of Participants with Antibodies to Guselkumab or Golimumab | Up to Week 36
  Percentage of participants with antibodies to guselkumab or golimumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (81):
- United States (19):
  - Arizona Arthritis and Rheumatology Research PLLC, Phoenix, Arizona
  - Unity Health-White County Medical Center, Searcy, Arkansas
  - HARAC Research Corp, Avon Park, Florida
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Omega Research Consultants, DeBary, Florida
  - South Coast Research Center, Miami, Florida
  - Advanced Clinical Research of Orlando, Ocoee, Florida
  - Millennium Research, Ormond Beach, Florida
  - Atlanta Research Center for Rheumatology, Marietta, Georgia
  - Great Lakes Center of Rheumatology, Lansing, Michigan
  - Clinvest, Springfield, Missouri
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - NYU School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Jacobi Medical Center, The Bronx, New York
  - STAT Research, Inc., Vandalia, Ohio
  - Trinity Universal Research Associates, LLC, Plano, Texas
  - DM Clinical Research, Tomball, Texas
  - Swedish Medical Center, Seattle, Washington
- Denmark (5):
  - Frederiksberg Hospital, Frederiksberg
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Køge Sygehus Region Sjaelland, Køge
  - Silkeborg Hospital, Silkeborg
  - Vejle Sygehus, Vejle
- France (3):
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Larrey CHU de Toulouse, Toulouse
  - CHU Trousseau - Service de Rhumatologie, Tours
- Hungary (4):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Bekes Varmegyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Complex Rendelo Med Zrt, Székesfehérvár
  - Vital Medical Center, Veszprém
- Italy (9):
  - Azienda Ospedaliero-Universitaria di Cagliari, Cagliari
  - Centro Specialistico Ortopedico Traumatologico Gaetano Pini CTO, Milan
  - Ospedale San Raffaele, Milan
  - IRCCS Policlinico San Matteo, Università degli studi di Pavi, Pavia
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - A.O.U.Policlinico Tor Vergata, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Università Campus Biomedico di Roma, Rome
  - AO Ordine Mauriziano, Torino
- Poland (7):
  - Centrum Kliniczno Badawcze, Elblag
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - NZOZ Lecznica MAK MED S C, Nadarzyn
  - Centrum Medyczne, Poznan
  - Medycyna Kliniczna, Warsaw
  - Centrum Medyczne AMED Targowek, Warsaw
  - WroMedica I Bielicka A Strzalkowska s c, Wroclaw
- Russia (11):
  - Kemerovo State Medical University, Kemerovo
  - LLL Medical Center Revma-Med, Kemerovo
  - LLC Family Outpatient Clinic # 4, Korolyov
  - GBUZ of Moscow Region 'Moscow Region SRI n.a. Vladimirskyi', Moscow
  - Orenburg State Medical Academy, Orenburg
  - Rostov Regional Clinical Dermatovenerological Dispensary, Rostov
  - Ryazan Regional Clinical Dermatovenerological Dispensary, Ryazan
  - X7 Clinical Research Company Limited, Saint Petersburg
  - Smolensk regional hospital on Smolensk railway station, Smolensk
  - Republican Clinical Hospital - G.G. Kuvatov, Ufa
  - Clinical Hospital #3, Yaroslavl
- Spain (10):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Univ. Germans Trias I Pujol, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. 12 de Octubre, Madrid
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Infanta Luisa, Seville
  - Hosp. Ntra. Sra. de Valme, Seville
- Sweden (2):
  - Skanes universitetssjukhus, Malmo
  - Karolinska Universitetssjukhuset Solna, Solna
- Ukraine (11):
  - State Institution Institute of therapy named after L.T.Malaya AMS Ukraine, Kharkiv
  - Municipal Institution Regional hospital-center of emergency care and disasters medicine, Kharkiv
  - Medical Research and Practice Center Medbud of the Public Joint Stock Holding Company Kyivmiskbud, Kyiv
  - Kyiv Railway Clinical Hospital #2 Of Branch 'Health Center' Of The Company 'Ukrainian Railway', Kyiv
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - Municipal Non-Profit Enterprise of Kyiv Regional Council 'Kyiv regional Clinical Hospital', Kyiv
  - ME Poltava Regional Clinical Hospital named after M.V. Sklifosovsky of Poltava Regional Consuil, Poltava
  - Municipal institution of Tepnopil Regional Council 'Ternopil University Hospital', Ternopil
  - MNCE Zakarpatska Regional Clinical Hospital named after A Novak of Zakarpatska Regional Council, Uzhhorod
  - Health Clinic Limited Liability Company, Vinnytsia
  - Medical Center LLC 'Modern Clinic', Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency